CLINICAL TRIAL: NCT01788007
Title: A Randomized, Double Blind, Placebo Controlled, Parallel Design, Multiple Site, Clinical Study to Evaluate the Bioequivalence of Two Imiquimod Cream 3.75% Formulations in Patients With Actinic Keratosis.
Brief Title: Clinical Study to Evaluate the Bioequivalence of Two Imiquimod Cream 3.75% Formulations in Patients With Actinic Keratosis.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMQC 1220
Record Dates: First submitted 2013-02-07; First posted 2013-02-11 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Actinic Keratosis
Keywords: Actinic Keratosis; Imiquimod Topical Cream 3.75%; Zyclara® (imiquimod) Topical Cream 3.75%
MeSH Terms: conditions — Keratosis, Actinic | interventions — Imiquimod

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Imiquimod Topical Cream 3.75% (Experimental): Imiquimod Topical Cream 3.75% (Taro Pharmaceutical Industries Ltd.)
  Interventions: Drug: Imiquimod Topical Cream 3.75%
- Vehicle Topical Cream (Placebo Comparator): Vehicle Topical Cream (Taro Pharmaceutical Industries Ltd.)
  Interventions: Drug: Vehicle Topical Cream
- Zyclara® (imiquimod) Topical Cream 3.75% (Active Comparator): Zyclara® (imiquimod) Topical Cream 3.75% (Medicis Pharmaceutical Co.)
  Interventions: Drug: Zyclara® (imiquimod) Topical Cream 3.75%

INTERVENTIONS:
Drug: Imiquimod Topical Cream 3.75% — Imiquimod Topical Cream 3.75% (Taro Pharmaceutical Industries Ltd.) applied once daily for two 14 day treatment cycles separated by a 14 day no treatment period.
  Arms: Imiquimod Topical Cream 3.75%
Drug: Zyclara® (imiquimod) Topical Cream 3.75% — Zyclara® (imiquimod) Topical Cream 3.75% (Medicis Pharmaceutical Co.) applied once daily for two 14 day treatment cycles separated by a 14 day no treatment period.
  Arms: Zyclara® (imiquimod) Topical Cream 3.75%
Drug: Vehicle Topical Cream — Vehicle Topical Cream (Taro Pharmaceutical Industries Ltd.) applied once daily for two 14 day treatment cycles separated by a 14 day no treatment period.
  Arms: Vehicle Topical Cream

SUMMARY:
The objective of this study is to compare the relative efficacy and safety of the test formulation Imiquimod 3.75% Topical Cream to the marketed formulation Zyclara® (imiquimod) 3.75% Topical Cream in the treatment of actinic keratosis. Both the test and reference formulations will also be compared to a placebo cream to test for superiority.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form.
* Immunocompetent male or non-pregnant, non-lactating female at least 18 years of age.
* Diagnosis of actinic keratosis with at least 5 and no more than 20 clinically typical, visible or palpable actinic keratosis lesions, each at least 4 mm in diameter, in an area that exceeds 25 cm2 on either the face (excluding ear) or balding scalp (but not both.)
* Women either must be 1 year post-menopausal, surgically sterile, or if they are of child-bearing potential, they must: a) have been using systemic birth control, intrauterine device, or Norplant for at least 28 days prior to the start of treatment period, or used barrier methods consistently, at least 14 days before study cream administration; b) had a normal menstrual cycle for the month prior to the start of treatment; c) have a negative urine pregnancy test result upon entry into the study; d) agree to use a medically accepted form of birth control throughout the study period.
* Free from any systemic or dermatologic disorder that, in the opinion of the Investigator, will interfere with the study results or increase the risk of adverse events.
* Any skin type or race, providing the skin pigmentation will allow discernment of erythema.
* Willingness and capability to cooperate to the extent and degree required by the protocol.

Exclusion Criteria:

* Presence of atopic dermatitis, basal cell carcinoma, squamous cell carcinoma, eczema, psoriasis, rosacea, sunburn or other possible confounding skin conditions on the face or bald scalp.
* Use within six months prior to baseline on the face or bald scalp of chemical peel, dermabrasion, laser abrasion, psoralen plus ultraviolet A therapy, or ultra violet B therapy.
* Use within one month prior to baseline on the face or bald scalp of cryodestruction or chemodestruction, curettage, photodynamic therapy, surgical excision, topical 5-fluorouracil, topical corticosteroids, topical diclofenac, topical imiquimod, topical retinoids or other treatments for actinic keratosis including glycolic acids or over-the-counter products containing retinol, alpha or beta hydroxy acids.
* Use within one month prior to baseline of immunomodulators or immunosuppressive therapies, interferon, oral corticosteroids or cytotoxic drugs.
* Known allergies to imiquimod or any excipients to the test or reference creams.
* Receiving 5-fluorouracil or other systemic cancer chemotherapy within 6 months prior to study entry.
* Any condition, medical, psychological, or social, that, in the Investigator's opinion, would interfere with participation in the study.
* Women who are pregnant or planning pregnancy or lactating during the study.
* Participation in any investigational drug study within 30 days of enrollment or previous participation in this study.
* Employees or family members of employees of the research center or Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 443 (Actual)
Dates: Start 2013-01; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Treatment success | Week 14 (8 weeks after completion of treatment)
  Treatment success will be defined by the proportion of patients in the per protocol population with 100% clearance of all actinic keratosis lesions within the treatment area at study week 14 (8 weeks after completion of treatment.)

SECONDARY OUTCOMES:
Superiority to placebo | Week 14 (8 weeks after completion of treatment)
  The modified intent-to-treat population and last observation carried forward will be used to evaluate the superiority of both the test and reference product to placebo for the proportion of patients showing 100% clearance of actinic keratosis lesions at week 14 (8 weeks after completion of treatment.)